CLINICAL TRIAL: NCT01165125
Title: A Double-blind, Randomized, Placebo-controlled, Repeat Dose, 2-way Crossover Drug Interaction Study to Investigate the Pharmacokinetic and Pharmacodynamic Effects Following Administration of Fluticasone Furoate/GW642444M Inhalation Powder With Ketoconazole
Brief Title: A Drug Interaction Study With Fluticasone Furoate/GW642444 Inhalation Powder and Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 105548
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: pharmacodynamics; drug interaction; ketoconazole; pharmacokinetics; Fluticasone furoate; GW642444
MeSH Terms: conditions — Asthma | interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/GW642444 and keto (Other): Ketoconazole (400mcg) administered on Days 1-11, with co-administration of fFF / GW642444 (200mcg/25mcg) on Days 5-11
  Interventions: Drug: FF / GW642444; Drug: ketoconazole
- Ketoconazole Placebo to match & FF/GW642444 (Other): ketoconazole placebo to match administered on days 1-11. FF/GW642444 (200mcg/25mcg) co-administered on Days 5-11
  Interventions: Drug: FF / GW642444; Drug: ketoconazole (placebo to match)

INTERVENTIONS:
Drug: FF / GW642444 — 200mcg/25mcg Novel DPI
Drug: ketoconazole — 400mcg overencapsulated tablets
  Arms: FF/GW642444 and keto
Drug: ketoconazole (placebo to match) — placebo to match overencapsulated tablets
  Arms: Ketoconazole Placebo to match & FF/GW642444

SUMMARY:
A randomized two-way crossover study to determine whether concomitant administration of CYP P450 3A4 inhibitor ketoconazole and fluticasone furoate/GW642444M combination significantly increases the systemic effects and exposure to repeat dose fluticasone furoate and/or GW642444 in healthy subjects. Key assessments will include blood potassium, heart rate, blood pressure, QTc, serum cortisol and pharmacokinetic parameters, and safety including vital signs, ECGs, adverse event monitoring and laboratory safety tests, including blood glucose.

DETAILED DESCRIPTION:
This will be a single centre, randomized, double-blind (with respect to ketoconazole), two-way cross-over study in healthy male and female subjects. Subjects will attend for a screening visit within 28 days prior to the first treatment period. There will be two study periods, each consisting of 14 days. Ketoconazole or matching placebo will be administered for 11 days with fluticasone furoate/GW642444M inhalation powder co-administered on Days 5-11. During each period subjects will be required to report to the unit on Day -1 and will remain there until 1 hour post-dosing with ketoconazole or placebo on Day 1. Subjects will return to the unit on the mornings of Day 2 to Day 4 for dosing with ketoconazole or placebo. Subjects will then return on the evening of Day 4 and leave the unit on the morning of Day 6 (2 nights). Subjects will return to the unit on the mornings of Day 7 to Day 10 for dosing and pre-fluticasone furoate/GW642444M dose safety assessments. Subjects will return on the evening of Day 10 and leave the unit on the morning of Day 12 (2 nights). Subjects will make two outpatient visits, one in the evening on Day 12 and one in the morning on Day 13, to complete a few study related procedures. The two treatment periods will be separated by a washout of at least 7 days and no more than 14 days. Pharmacodynamic profiles for potassium, heart rate, QTc, blood pressure and serum cortisol will be taken on Day 11 with fluticasone furoate and GW642444 pharmacokinetic profiles on Days 5 and 11. Safety assessments will include vital signs, ECGs, adverse event monitoring and laboratory safety tests, plus blood glucose and blood potassium profiles on Day 5.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between 18 and 64 years of age inclusive
2. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.
3. Body mass index within range of 18.5-29.0 kg/m2 inclusive.
4. Subjects who are current non-smokers, who have not used any tobacco products in the 12 month period preceding the screening visit, and have a pack history of </= 5 pack years.
5. AST, ALT, alkaline phosphatase and bilirubin </= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
6. No significant abnormality on 12-lead ECG at screening, including the following specific requirements:

   * QTcF < 450 msec
7. No clinically significant abnormality on the Holter ECG at screening.
8. FEV1 >/= 85% predicted at screening.
9. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
10. Able to satisfactorily use the dry powder inhaler.

Exclusion Criteria:

1. As a result of medical interview, physical examination or screening investigations, the principal investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age.
2. The subject has any history of breathing problems in adult life (i.e. history of asthmatic symptomatology).
3. Pregnant females as determined by positive serum hCG test at screening or by positive serum/urine hCG test prior to dosing.
4. Lactating females.
5. The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
6. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
7. Subjects who have suffered a lower respiratory tract infection within 4 weeks of the screening visit.
8. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
9. Any adverse reaction including immediate or delayed hypersensitivity to any beta-agonist, sympathomimetic drug, or any intranasal, inhaled or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the new powder inhaler (ie lactose or magnesium stearate)
10. History of milk protein allergy.
11. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
12. The subject has taken oral corticosteroids less than 8 weeks before the screening visit.
13. The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
14. History of alcohol/drug abuse or dependence within 12 months of the study. Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females).
15. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
16. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
17. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months of the start of the trial.
18. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
19. The subject has tested positive for HIV antibodies.
20. A positive pre-study urine drug screen or when randomly tested during the study.
21. Positive carbon monoxide (CO) or alcohol breath test at screening or on admission to the Unit.
22. Consumption of seville oranges, pomelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication.
23. Unwillingness or inability to follow the procedures outlined in the protocol.
24. Subject is mentally or legally incapacitated.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2010-08-28 (Actual); Study Completion 2010-08-28 (Actual)

PRIMARY OUTCOMES:
Maximum heart rate (0-4 hours) and minimum blood potassium level (0-4 hours) on the morning of Day 11 | Day 11
Weighted mean serum cortisol (0-24 hours) on Day 11. | Day 11

SECONDARY OUTCOMES:
Minimum diastolic blood pressure (0-4 hours), maximum systolic blood pressure (0-4 hours) and maximum QTcF (0-4 hours) on the morning of Day 11 | Day 11
Fluticasone furoate and GW642444 pharmacokinetics (AUC(0-t), AUC(0-24), Cmax, tmax) on Day 5 and 11 | day 11
Reported adverse events | 2 months
12-lead ECG and clinical laboratory data and maximum heart rate (0-4 hours) maximum QTc (0-4 hours) and minimum blood potassium and blood glucose levels (0-4 hours) on the morning of Day 5. | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kempsford R, Allen A, Bal J, Rubin D, Tombs L. The effect of ketoconazole on the pharmacokinetics and pharmacodynamics of inhaled fluticasone furoate and vilanterol trifenatate in healthy subjects. Br J Clin Pharmacol. 2013 Jun;75(6):1478-87. doi: 10.1111/bcp.12019. PMID 23116485
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 105548 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/105548?search=study&study_ids=105548#rs
- Available data/document: Dataset Specification: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105548 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register